CLINICAL TRIAL: NCT03719183
Title: Comparison of Diagnostic Yield Among Multiplex Fluorescent in Situ Hybridization, Fluorescent in Situ Hybridization Probe Panel and Conventional Cytogenetic Studies in Acute Myeloid Leukemia
Brief Title: Comparison of Diagnostic Yield Among M-FISH, FISH Probe Panel and Conventional Cytogenetic Analysis in AML
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Collaborators: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Ahmed Makboul Ahmed Makboul, Assistant Lecturer, Assiut University
Other Study IDs: AssiutU-SECI-Cytogenetic 100
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: M-FISH, FISH, AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Karyotyping; In Situ Hybridization; In Situ Hybridization, Fluorescence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral blood or Bone marrow aspiration samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Myeloid Leukemia (AML) group: Patients who are diagnosed as Acute Myeloid Leukemia based on peripheral blood, bone marrow aspiration and immunophenotyping and fulfill WHO criteria for diagnosis.
  Fluorescent in Situ Hybridization (FISH) Panels for AML, Multiplex FISH (M-FISH) and Conventional Cytogenetics Studies will be performed for AML patients.
  Interventions: Diagnostic Test: Conventional Cytogenetics Studies; Diagnostic Test: Fluorescent in Situ Hybridization (FISH) Panels; Diagnostic Test: Multiplex FISH (M-FISH)

INTERVENTIONS:
Diagnostic Test: Conventional Cytogenetics Studies — Metaphase cytogenetic studies will be performed in all cases according to standard methods. Chromosome preparations will be G-banded using trypsin and Giemsa, and karyotypes will be described according to the International System for Human Cytogenetic Nomenclature (ISCN) 2016.
  Other Names: Karyotyping
Diagnostic Test: Fluorescent in Situ Hybridization (FISH) Panels — AML Panel includes:
  * t(8;21) (RUNX1-RUNX1T1).
  * inv(16), t(16;16) (CBFB-MYH11).
  * t(9;22) (BCR-ABL).
  * 11q23 KMT2A rearrangements.
  * inv(3) MECOM rearrangements.
  * DEK-NUP214 rearrangements.
  * Del(5q) Deletion
  * Del(7q) Deletion
  Acute Promyelocytic Leukemia panel includes:
  * t(15;17) (PML-RARA).
  * 17q RARA rearrangements
Diagnostic Test: Multiplex FISH (M-FISH) — 24-color karyotyping

SUMMARY:
Conventional cytogenetic studies have been the gold standard for more than five decades for detecting genetic alterations that are greater than 10 Mb (mega base pairs) in size. Conventional cytogenetic studies have paved the way in identifying specific chromosomal aberrations associated with clinically and morphologically definitive subsets of hematological neoplasms.

Fluorescence in situ hybridization (FISH) has become a reliable and rapid complementary test in targeting critical genetic events associated with diagnostics and prognosis in hematological neoplasms.

In the current health care environment, which increasingly focuses on value and efficiency, it is critical for pathologists and clinicians to effectively navigate this environment and judiciously incorporate these high-complexity and expensive techniques into routine patient care. While conventional karyotyping provides a comprehensive view of the genome, FISH can detect cryptic or submicroscopic genetic abnormalities and identify recurrent genetic abnormalities in nondividing cells. As a consequence, it is commonly extrapolated that FISH will improve the sensitivity of detecting all genetic abnormalities compared with conventional karyotyping analysis. This assumption has then been translated in clinical practice to having clinicians and pathologists routinely ordering both conventional karyotyping and FISH studies in patients with hematological neoplasms. Depending on how comprehensive the FISH panel is, the cost for this testing may be quite expensive, and its additive value remains questionable.

It is common practice for laboratories to use FISH panels in conjunction with karyotyping both in diagnostic specimens and during follow-up to monitor response to therapy.

Multiplex FISH (M-FISH) represents one of the most significant developments in molecular cytogenetics of the past decade. In tumor and leukemia cytogenetics, two groups have been targeted by M-FISH to identify cryptic chromosome rearrangements not detectable by conventional cytogenetic studies: those with an apparently normal karyotype (suspected of harboring small rearrangements not detectable by conventional cytogenetics) and those with a complex aberrant karyotype (which are difficult to karyotype accurately due to the sheer number of aberrations).

DETAILED DESCRIPTION:
Neoplastic hematology is at the forefront of personal¬ized medicine. The World Health Organization (WHO) classification incorporates genetic data with microscopic, immunophenotypic, and clini¬cal findings and categorizes hematologic neoplasms into clinically and biologically distinct categories. This system guides diagnosis, prognosis and therapeutic choices, which has become increasingly important with emerging targeted therapies for lymphoma and leukemia. However, laboratory tests for hematologic neoplasms are of high complexity and are generally quite costly.

The initial assessment of many hematologic neoplasms includes morphological, histological, immunophenotypic (flow cytometric and/or immunohistochemical), and conventional cytogenetic studies. Data obtained from cytogenetic analysis can be pathognomonic for specific leukemias in the WHO classification (for example, acute myeloid leukemia (AML) with recurrent cytogenetic abnormalities and chronic myelogenous leukemia (CML)) and are likely to assume a greater role in defining specific categories in further classifications.

Conventional cytogenetic studies have been the gold standard for more than five decades for detecting genetic alterations that are greater than 10 Mb (mega base pairs) in size. They have paved the way in identifying specific chromosomal aberrations associated with clinically and morphologically definitive subsets of hematological neoplasms.

Fluorescent in situ hybridization (FISH) has become a reliable and rapid complementary test in targeting critical genetic events associated with diagnostics and prognosis in hematological neoplasms. FISH has addressed the issues with conventional cytogenetic studies by targeting interphase cells in addition to metaphases. It has become clear that FISH studies may also be an integral component of the diagnostic evaluation, particularly where the abnormality is "cryptic" i.e. not evident by conventional cytogenetic studies.

Although complementary FISH testing increases the overall detection of aberrations, its benefit is not uniform across all types of hematological neoplasms. This is because FISH probes are restricted to the detection of only specific abnormalities and genetic alterations beyond the scope of the FISH probes would therefore be completely missed.

It is common practice for laboratories to use FISH probe panels in conjunction with karyotyping both in diagnostic specimens and during follow-up to monitor response to therapy. FISH is targeted toward specific abnormalities, and results can be evaluated in an automated fashion on interphase nuclei, allowing for examination of more cells than conventional cytogenetic studies. FISH has higher analytic and, in certain circumstances, higher clinical sensitivity compared with conventional cytogenetic studies. The usage of FISH probe panels in aiding diagnosis or in monitoring follow-up samples of hematologic neoplasms is critical.

The Eastern Collaborative Oncology Group (ECOG) compared conventional cytogenetic studies and FISH in AML patients and found that a probe panel to detect monosomy 5/deletion 5q, monosomy 7/deletion 7q, trisomy 8, t(8;21), t(9;22), MLL rearrangements with various partners, t(15;17), and inv(16)/t(16;16), had a concordance between 98% and 100%. On the other hand, He et al study demonstrates the limited value of FISH testing in adult AML in the setting of an adequate karyotyping study.

Despite of many significant technological advances made in recent years in the area of clinical genetic testing, conventional cytogenetic studies and routine FISH studies remain important laboratory testing tools available for evaluating hematologic neoplasms. Usually these two testing methods complement each other and often FISH serves to clarify and better define cytogenetic results. Therefore, there is a very strong expectation that cytogenetic and FISH results should confirm each other in spite of cases that appear to be exceptions. When conflicting results occur by these two testing methods on the same specimen, clinical laboratories are challenged to offer explanations based on empirical data beyond simply stating that it was or was not due to laboratory error.

Multiplex FISH (M-FISH) represents one of the most significant developments in molecular cytogenetics of the past decade. In tumor and leukemia cytogenetics, two groups have been targeted by M-FISH to identify cryptic chromosome rearrangements not detectable by conventional cytogenetic studies: those with an apparently normal karyotype (suspected of harboring small rearrangements not detectable by conventional cytogenetics) and those with a complex aberrant karyotype (which are difficult to karyotype accurately due to the sheer number of aberrations).

Zhang et al. used spectral karyotype (SKY) to re-evaluate the karyotypes of AML cases reported as normal by G-banding. This resulted in the identification of one case of t(11;19)(q23;p13), a subtle but recognized cytogenetic abnormality, and a minor clone containing monosomy for chromosome 7 in another case. In a similar study, Mohr et al. compared SKY to conventional karyotyping in patients with AML or MDS with normal karyotypes. No abnormalities were identified.

With the lack of an evidence-based standardized algorithmic approach, misuse and overutilization of laboratory tests are common and result in increased health care costs and patient care complexity. In the current health care environment, which increasingly focuses on value and efficiency, it is critical for pathologists and clinicians to incorporate high-complexity and expensive techniques into routine patient care. While conventional cytogenetic studies provide a comprehensive view of the genome, FISH probe panel can detect cryptic or submicroscopic genetic abnormalities and identify recurrent genetic abnormalities in nondividing cells. M-FISH can identify cryptic chromosome rearrangements that are not detected by conventional cytogenetic studies. As a consequence, it is commonly extrapolated that FISH will improve the sensitivity of detecting all genetic abnormalities compared with conventional cytogenetic studies. This assumption has then been translated in clinical practice to having clinicians and pathologists routinely ordering both conventional cytogenetic studies and FISH studies in patients with hematological neoplasms. Depending on how comprehensive the FISH probe panel is, the cost for this testing may be quite expensive, and its additive value remains questionable.

ELIGIBILITY:
Inclusion criteria:

1. Patients with newly diagnosed acute myeloid leukemia.
2. Age group: patients more than 18 years old.

Exclusion criteria:

1. Patients less than 18 years old.
2. Patients with other types of hematologic neoplasms.
3. Relapsed patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed AML patients.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of cytogenetic profile of AML patients in South Egypt | 2 years
  Study the hematological and cytogenetic profile of AML patients in a tertiary center in Egypt
Comparing Diagnostic Yield among Multiplex Fluorescent in situ hybridization, fluorescent in situ hybridization probe panel and conventional cytogenetic analysis in newly diagnosed patients with AML. | 2 years
  Compare M-FISH, karyotyping and FISH probe panel in AML patients in a limited resource institute

SECONDARY OUTCOMES:
Correlation between cytogenetic results and demographic, clinical and hematological data of AML patients | 2 years
  Correlating cytogenetic results and demographic and clinicopathological data in AML patients

CONTACTS AND LOCATIONS:
Overall Officials: Eman Mosaad, MD, Study Director — South Egypt Cancer Institute
Locations (1):
- South Egypt Cancer Institute, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ashok V, Ranganathan R, Chander S, Damodar S, Bhat S, S NK, A SK, Jadav SS, Rajashekaraiah M, T S S. Comparison of Diagnostic Yield of a FISH Panel Against Conventional Cytogenetic Studies for Hematological Malignancies: A South Indian Referral Laboratory Analysis Of 201 Cases. Asian Pac J Cancer Prev. 2017 Dec 29;18(12):3457-3464. doi: 10.22034/APJCP.2017.18.12.3457. PMID 29286619
- [Background] Cantu ES, Dong H, Forsyth DR, Espinoza FP, Papenhausen PR. Discrepant Cytogenetic and Interphase Fluorescence In Situ Hybridization (I-FISH) Results from Bone Marrow Specimens of Patients with Hematologic Neoplasms. Ann Clin Lab Sci. 2018 May;48(3):264-272. PMID 29970427
- [Background] He R, Wiktor AE, Hanson CA, Ketterling RP, Kurtin PJ, Van Dyke DL, Litzow MR, Howard MT, Reichard KK. Conventional karyotyping and fluorescence in situ hybridization: an effective utilization strategy in diagnostic adult acute myeloid leukemia. Am J Clin Pathol. 2015 Jun;143(6):873-8. doi: 10.1309/AJCPP6LVMQG4LNCK. PMID 25972330
- [Background] Kearney L. Multiplex-FISH (M-FISH): technique, developments and applications. Cytogenet Genome Res. 2006;114(3-4):189-98. doi: 10.1159/000094202. PMID 16954655
- [Background] Kokate P, Dalvi R, Koppaka N, Mandava S. Prognostic classification of MDS is improved by the inclusion of FISH panel testing with conventional cytogenetics. Cancer Genet. 2017 Oct;216-217:120-127. doi: 10.1016/j.cancergen.2017.05.004. Epub 2017 Aug 16. PMID 29025586
- [Background] Mohr B, Bornhauser M, Thiede C, Schakel U, Schaich M, Illmer T, Pascheberg U, Ehninger G. Comparison of spectral karyotyping and conventional cytogenetics in 39 patients with acute myeloid leukemia and myelodysplastic syndrome. Leukemia. 2000 Jun;14(6):1031-8. doi: 10.1038/sj.leu.2401775. PMID 10865969
- [Background] Peterson JF, Aggarwal N, Smith CA, Gollin SM, Surti U, Rajkovic A, Swerdlow SH, Yatsenko SA. Integration of microarray analysis into the clinical diagnosis of hematological malignancies: How much can we improve cytogenetic testing? Oncotarget. 2015 Aug 7;6(22):18845-62. doi: 10.18632/oncotarget.4586. PMID 26299921
- [Background] Sreekantaiah C. FISH panels for hematologic malignancies. Cytogenet Genome Res. 2007;118(2-4):284-96. doi: 10.1159/000108312. PMID 18000382
- [Background] Vance GH, Kim H, Hicks GA, Cherry AM, Higgins R, Hulshizer RL, Tallman MS, Fernandez HF, Dewald GW. Utility of interphase FISH to stratify patients into cytogenetic risk categories at diagnosis of AML in an Eastern Cooperative Oncology Group (ECOG) clinical trial (E1900). Leuk Res. 2007 May;31(5):605-9. doi: 10.1016/j.leukres.2006.07.026. Epub 2006 Sep 22. PMID 16996130
- [Background] Wheeler FC, Kim AS, Mosse CA, Shaver AC, Yenamandra A, Seegmiller AC. Limited Utility of Fluorescence In Situ Hybridization for Recurrent Abnormalities in Acute Myeloid Leukemia at Diagnosis and Follow-up. Am J Clin Pathol. 2018 Mar 29;149(5):418-424. doi: 10.1093/ajcp/aqy002. PMID 29538617
- [Background] Wolff DJ, Bagg A, Cooley LD, Dewald GW, Hirsch BA, Jacky PB, Rao KW, Rao PN; Association for Molecular Pathology Clinical Practice Committee; American College of Medical Genetics Laboratory Quality Assurance Committee. Guidance for fluorescence in situ hybridization testing in hematologic disorders. J Mol Diagn. 2007 Apr;9(2):134-43. doi: 10.2353/jmoldx.2007.060128. PMID 17384204
- [Background] Zhang FF, Murata-Collins JL, Gaytan P, Forman SJ, Kopecky KJ, Willman CL, Appelbaum FR, Slovak ML. Twenty-four-color spectral karyotyping reveals chromosome aberrations in cytogenetically normal acute myeloid leukemia. Genes Chromosomes Cancer. 2000 Jul;28(3):318-28. doi: 10.1002/1098-2264(200007)28:33.0.co;2-m. PMID 10862038